CLINICAL TRIAL: NCT03131661
Title: A Prospective, Observational Study, in Patients With a Newly Confirmed Diagnosis of Spondyloarthritis (SpA) According to ASAS Criteria, naïve to Conventional (cDMARDs), Targeted (tsDMARDs) and Biological DMARDs (bDMARDs) - SIRENA Study (Spondyloarthritis Italian Registry: Evidence From a National Pathway)
Brief Title: A Study in Participants With a Newly Confirmed Diagnosis of Spondyloarthritis (SpA) Who Are New to Conventional, Targeted and Biological DMARDs
Acronym: SIRENA
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108297; CNTO1275PSA4006 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Spondyloarthritis, Axial and Peripheral
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SpA with DMARDs: Participants with first diagnosis or confirmed diagnosis of Spondyloarthritis (SpA) and naïve to conventional, targeted or biological Disease modifying anti-rheumatic drugs (DMARDs) will be observed in order to describe SpA characteristics and pattern of clinical presentation.

SUMMARY:
The purpose of this Italian multicenter study is to collect prospective clinical data in participants with first diagnosis or confirmation diagnosis of Spondyloarthritis (SpA), according to Assessment of Spondyloarthritis classification (ASAS) criteria, in order to describe SpA characteristics and pattern of clinical presentation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a first or confirmed diagnosis of Spondyloarthritis (SpA) according to Assessment of Spondyloarthritis classification (ASAS) criteria
* Participants must be naïve to conventional, targeted and biological Disease modifying anti-rheumatic drugs (DMARDs) treatment
* Participants must understand the purpose of the study
* Participants must sign a participation agreement/ Informed Consent Form (ICF) allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

* Participants who already started conventional, targeted and biological DMARDs treatment for SpA
* Participants who participate to an investigational study in the last 30 days
* Participants unwilling or unable to participate in long-term, 24 months, data collection
* Participants unwilling or unable to fill in the Participant-reported outcome (PRO) foreseen by the protocol
* Participants unwilling or unable to sign the informed consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include outpatients with first diagnosis or confirmed diagnosis of Spondyloarthritis (SpA) and naïve to conventional, targeted or biological Disease modifying anti-rheumatic drugs (DMARDs) prescribed for SpA.
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic Delay | Baseline (Month 0)
  Time of diagnostic delay, defined as the time in months from first symptoms to diagnosis, and reasons for this delay.
Prevalence of Axial Versus Peripheral Manifestations According to Assessment of Spondyloarthritis Classification (ASAS) Criteria | Up to visit 5 (Approximately 24 months)
  The ASAS criteria distinguish axial from peripheral SpA. ASAS criteria for axial SpA: chronic back pain (>=3 months) with onset at age <45 years, and include imaging and clinical arm. Imaging criteria: must have sacroiliitis visible on either pelvic radiograph (representing the Ankylosing Spondylitis subgroup) or active inflammation detected by Magnetic Resonance Imagining (MRI) of the sacroiliac joints, and at least one other feature of SpA. Clinical criteria: should be Human Leukocyte Antigen (HLA) B27 positive and have at least two other SpA associated features. ASAS criteria for peripheral manifestations: must have arthritis, dactylitis or enthesitis in combination with either at least one of psoriasis, inflammatory bowel disease, uveitis, preceding genitourinary or gastro intestinal infection, HLA B27 positivity or sacroiliitis, or with two or more of arthritis, dactylitis, enthesitis, inflammatory back pain (at any time in the participant's history) or a family history of SpA.
Effectiveness for cDMARDs, tDMARDs, bDMARDs: Assessed by ASDAS Score | Up to visit 5 (Approximately 24 months)
  The ASDAS is composite score based on the calculation of 5 disease activities: 4 are participant's reported outcomes (back pain, duration of morning stiffness, participant global and peripheral pain/swelling) and one serologic inflammation marker (C-reactive protein [CRP]). The score is the sum of the 5 items with different specified weights, with a minimum of 0 and no upper limit. Thus this index can reflect both long term disease activity and acute phase status. There are 2 cut-offs in score to show: a) the 4 states of disease activity: inactive disease (less than [<] 1.3), moderate disease activity (1.3-2.1), high disease activity (2.1-3.5) and very high disease activity (greater than [>] 3.5). b) effectiveness of the treatment, two validated cut-offs were developed: a change of 1.1-2.0 (clinically important improvement) and a change >2.0 (major improvement).
Effectiveness for cDMARDs, tDMARDs, bDMARDs: Assessed by BASMI Score | Up to visit 5 (Approximately 24 months)
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) is an index for measuring the mobility of the axial skeleton in participant affected by ankylosing spondylitis (AS). This index consists of 5 clinical measurements, including lumber side flexion, tragus to wall distance, lumbar flexion, intermalleoar distance and cervical rotation. Individual scores are averaged to give a final score between 0 and 10. A higher BASMI10 score reflects more severe spinal mobility limitation.
Effectiveness for cDMARDs, tDMARDs, bDMARDs: Assessed by DAS28 Score | Up to visit 5 (Approximately 24 month)
  The Disease Activity and functional status assessment (DAS) 28 score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment of disease activity [visual analog scale: 0 = no disease activity to 100 = maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement. European League Against Rheumatism (EULAR) Good response: DAS28 less than or equal to (<=) 3.2 or a change from Baseline less than (<) -1.2. EULAR Moderate response: DAS28 greater than (>) 3.2 to <= 5.1 or a change from Baseline < -0.6 to greater than or equal to (>=) -1.2.
Effectiveness for cDMARDs, tDMARDs, bDMARDs: Assessed by Disease Activity Index for PsA (DAPSA) Score | Up to visit 5 (Approximately 24 months)
  The DAPSA score will be calculated by the data collection tool and is the sum of the following: Participant's assessment of pain on visual analog scale (VAS) (in centimeters), Participant's Global Assessment of Disease Activity on VAS, 66 and 68 joint counts for swelling and tenderness, respectively. Joints assessed include the distal interphalangeal (DIP), proximal interphalangeal (PIP), and metacarpophalangeal (MCP) joints of the hands; the wrist, elbow, shoulder, acromioclavicular, sternoclavicular, temporomandibular, hip (excluded for swelling), knee, ankle, and midtarsal joints; and the metatarsophalangeal and PIP joints of the feet. CRP level in milligrams per deciliters (mg/dL). Cutoff values for low and high disease activity are <= 18.5 and >= 45.1 points, 25 respectively, and for remission is <= 3.3 points.
Effectiveness for cDMARDs, tDMARDs, bDMARDs: Assessed by MDA | Up to visit 5 (Approximately 24 months)
  Minimal Disease Activity (MDA) is a state of disease activity deemed a useful target of treatment by both the participant and physician. The goal of the development of this instrument is to "treat to target" to achieve disease remission or low disease activity state. For a participant to achieve MDA, 5 of the following 7 criteria must be met: Tender joint count =<1; Swollen joint count =<1; Psoriasis Area and Severity Index (PASI) =<1 or Body surface area (BSA) =<3; Participant pain VAS =<15; Participant global activity VAS =<20; HAQ =<0.5; Tender enthesial points =<1.
Drug Retention for cDMARDs, tDMARDs and bDMARDs | Up to visit 5 (Approximately 24 months)
  Drug Retention is defined as the time in months in which participants maintain the same therapy.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to visit 5 (Approximately 24 months)
  An adverse event is any untoward medical occurrence in a clinical study that does not necessarily have a causal relationship with the investigational drug under study.

SECONDARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Score (ASDAS) C-reactive Protein (CRP) | Up to visit 5 (Approximately 24 month)
  The ASDAS is an index for measuring disease activity in participant affected by ankylosing spondylitis. The ASDAS-CRP is derived from back pain, duration of morning stiffness, general well being, C-reactive protein (CRP) and peripheral joint pain/swelling. Total score ranges from zero (reflecting no disease activity) with the upper end of the scale being determined by the level of CRP. The scores were categorized as follows : inactive disease (< 1.3), moderate (1.3 - < 2.1), high (2.1 - 3.5) and very high disease activity (> 3.5).
Bath Ankylosing Spondylitis Metrology Index (BASMI) 10 | Up to visit 5 (Approximately 24 month)
  The BASMI is an index for measuring the mobility of the axial skeleton in participant affected by ankylosing spondylitis. This index consists of 5 clinical measurements, including lumber side flexion, tragus to wall distance, lumbar flexion, intermalleoar distance and cervical rotation. Individual scores are averaged to give a final score between 0 and 10. A higher BASMI10 score reflects more severe spinal mobility limitation.
Disease Activity Score (DAS) 28 | Up to visit 5 (Approximately 24 month)
  The DAS 28 is a composite score derived from the following 4 measures. The index considers four parameters to obtain the total score: Count the number of swollen joints (out of the 28); Count the number of tender joints (out of the 28); C-reactive protein (CRP) expressed in milligram per milliLitre (mg/mL); Participant's Global Assessment of disease activity.
Disease Activity Index for Psoriatic Arthritis (DAPSA) | Up to visit 5 (Approximately 24 month)
  The DAPSA is a score used to measure disease activity in participant affected by psoriatic arthritis. It comprises: 68 tender and 66 swollen joints count; Participant global assessment of health; Participant pain Visual analogue scale (VAS); C-reactive protein level (milligram per deciLiter [mg/dl]).
Minimal Disease Activity (MDA) | Up to visit 5 (Approximately 24 month)
  The MDA is a state of disease activity deemed a useful target of treatment by both the participant and physician. For a participant to achieve MDA, 5 of the following 7 criteria must be met: Tender joint count less than or equal to (<=) 1; Swollen joint count <= 1; PASI <= 1 or BSA <= 3; Participant pain VAS <= 15; Participant global activity VAS <= 20; Health Assessment Questionnaire (HAQ) <= 0.5; Tender enthesial points <= 1.
Body Surface Area (BSA) | Up to visit 5 (Approximately 24 month)
  The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand (entire palmar surface or "handprint" which equates to approximately 1 % of total body surface area. The disease severity will be classified using the following categories: mild (BSA less than [<] 3 %), moderate (BSA from 3% to 10%), and severe (BSA more than [>] 10 %).
Bath Ankylosing Spondylitis Functional Index (BASFI) | Up to visit 5 (Approximately 24 month)
  The BASFI is used to define and monitor physical functioning in participants with ankylosing spondylitis. BASFI is composed by 10 items. Score range is 0-10, with 0 (easy), reflecting no functional impairments, and 10 (impossible), reflecting maximal impairment.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Up to visit 5 (Approximately 24 month)
  The BASDAI is used to measure participant reported disease activity in participants with ankylosing spondylitis. A numeric response scale (0-10) with "none" and "very severe" is used to answer. The final score ranges from 0 (no disease activity) to 10 (maximal disease activity). A cut off of 4 is used to define active disease.
Health Assessment Questionnaire - Disability Index (HAQ-DI) | Up to visit 5 (Approximately 24 month)
  The HAQ-DI is used to assess the physical functioning of the participant.The participant is required to indicate the degree of difficulty they have experienced, in each 8 items of the questionnaire, in the past week, in a 4 point scale. The responses in each functional area are: 0 = able to do with no difficulty; 1 = able to do with some difficulty; 2 = able to do with much difficulty; and 3 = unable to do. The 10 individual subscale scores are averaged to give a summary score. The range of the final calculates summary score is 0-3 where lower scores are indicative of better functioning and higher score reflects worse function. HAQ-DI scores of 0 to 1 generally represent mild to moderate functional difficulty, 1 to 2 represent moderate to severe functional difficulty, and 2 to 3 indicate severe to very severe limitations of physical function or disability.
Work Productivity and Activity Impairment Questionnaire (WPAI-SHP) | Up to visit 5 (Approximately 24 month)
  The WPAI is a validated, self administered questionnaire that assesses work and activity impairment during the past 7 days. The WPAI-SHP outcomes are expressed as impairment percentages; with higher numbers indicate greater impairment and less productivity, that is, worse outcomes.

OTHER OUTCOMES:
Number of Participants With 66/68 Swollen/Tender Joints Count | Up to 5 visits (approximately 24 months)
  Participant's swollen and tender joints 66/68 will be evaluated at each visit.
Physician Global Assessment of Participant (PhGA) Joints and Skin | Up to 5 visits (approximately 24 months)
  The PhGA, joint and skin, will be manually filled in by physician and will be documented using a VAS scale. PhGA VAS for pain ranges from "Quite" (0 millimeter [mm]) to "Very Severe" (100 mm); VAS for joint ranges from "No Inflammation" (0 mm) to "Very Severe" (100 mm); VAS for skin ranges from "Clear" (0 mm) to "Very Severe" (100 mm).
Number of Participants With Enthesitis | Up to 5 visits (approximately 24 months)
  The Maastricht Ankylosing Spondylitis Entheses Score (MASES) is a feasible index using to investigate the enthesitis. 13 specific and sensitive sites were examined and a dichotomous 0/1 score is used to value the grading of tenderness.
Number of Participants With Nail Lesions | Up to 5 visits (approximately 24 months)
  Number of participants with count of nail lesions will be presented.
Number of Participants With Dactylitis | Up to 5 visits (approximately 24 months)
  The total number of digits of the hands and feet (that is, 0 to 20) with dactylitis will be evaluated.
Number of Participants With Fibromyalgia | Up to 5 visits (approximately 24 months)
  Fibromyalgia is evaluated by American College of Rheumatology (ACR) 2010 criteria.
Number of Participants With Pain by Visual Analog Scale (VAS) | Up to 5 visits (approximately 24 months)
  The pain VAS is a self-administered assessment used to measure the average pain during the past week. The score ranges between 0 "No pain" to 0 "The Worst Possible Pain".
Number of Participants With Sleep Quality by VAS | Up to 5 visits (approximately 24 months)
  The Sleep Quality VAS questionnaire provides a measurement of quality of sleep experienced by the participant. This subjective method attempts to measure qualitative aspects of sleep and is easily administered. The score ranges from between 0 "Very Good" to 100 "Very Bad".
Participant's Global Assessment (PtGA) by VAS | Up to 5 visits (approximately 24 months)
  The PtGA by VAS measuring the overall way the disease affects the participants at a point in time. The score will be recorded as a single vertical mark on a 100 millimeter (mm) visual analogic scale (VAS), with 0 representing the lowest level of disease activity and 100 representing the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.
Locations (25):
- Italy (25):
  - ASST Spedali Civili Brescia, Brescia
  - Ospedale 'Antonio Cardarelli' di Campobasso - Azienda Sanitaria Regionale del Molise, Campobasso
  - P.O. Vittorio Emanuele Azienda Ospedaliero Universitaria 'Policlinico Vittorio Emanuele', Catania
  - AO di Catanzaro 'Pugliese Ciaccio', Catanzaro
  - Azienda Ospedaliera Mater Domini, Catanzaro
  - Ospedali Riuniti Foggia, Foggia
  - Ospedale La Colletta-Arenzano ASL3 Genovese, Genova
  - Ospedale San Raffaele, IRCCS, Milan
  - Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - P.O. 'Sant'Antonio', Padua
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera di Perugia Ospedale S.Maria della Misericordia, Perugia
  - Presidio Ospedaliero Pescara, Pescara
  - Ospedale San Carlo Di Potenza - Azienda Ospedaliera Regionale, Potenza
  - Policlinico Tor Vergata, Roma
  - Humanitas Hospital, Rozzano (MI)
  - Operative Unit of Rheumathology, Presidio Ospedaliero Vito Fazzi - Stabilimento Osp. A. Galateo, San Cesareo Di Lecce
  - Ospedale Busacca - Azienda Provinciale Sanitaria di Ragusa, Scicli (Ragusa)
  - Azienda Ospedaliera Universitaria Senese, Siena
  - A.O. Universitaria Ospedali Riuniti di Ancona, Torrette - Ancona
  - ASUI Santa Maria della Misericordia di Udine, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona

REFERENCES:
- [Derived] Favalli EG, Luchetti Gentiloni MM, Selmi C, Ramonda R, Grembiale RD, Dagna L, D'Angelo S, Gerli R, Foti R, Ciccia F, Guggino G, Franceschini F, Chimenti MS, Rossini M, Lubrano E, Frediani B, Marelli S, Zabotti A. The Impact of Sex on the Pattern and Clinical Response of Early Psoriatic Arthritis: Real-life Data from the Italian Prospective SIRENA Study. Rheumatol Ther. 2025 Oct;12(5):941-960. doi: 10.1007/s40744-025-00787-1. Epub 2025 Jul 25. PMID 40715761